CLINICAL TRIAL: NCT01272362
Title: Study of the Predictive Value of Airway Obstruction Reversibility on the Effectiveness of Indacaterol (Onbrez® Breezhaler ®) 150 mcg Once Daily in Patients With Moderate to Severe COPD
Brief Title: To Determine the Relationship Between Baseline Reversibility and the Efficacy of Indacaterol
Acronym: REVERBREZ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQAB149BFR01; 2010-022831-12 (EudraCT Number)
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Indacaterol; COPD; LABA; Reversibility
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

ARMS (1):
- Indacaterol (Experimental)
  Interventions: Drug: Indacaterol

INTERVENTIONS:
Drug: Indacaterol — Indacaterol 150 µg once-daily via single-dose dry powder inhaler

SUMMARY:
In this 5-months study, the response of patients to salbutamol at baseline will be compared with their response to treatment with indacaterol.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD (moderate-to-severe as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines, 2009) and:

  1. Post-bronchodilator FEV1 <80% and ≥30% of the predicted normal value
  2. Post-bronchodilator FEV1/FVC (forced vital capacity) <70%
* Smoking history of at least 10 pack-years

Exclusion Criteria:

* Patients who have had a COPD exacerbation in the 6 weeks prior to screening
* Patients who have had a respiratory tract infection within 4 weeks prior to screening
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular comorbid conditions

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 625 (Actual)
Dates: Start 2010-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Coefficient of correlation between FEV1 and reversibility | After 1 month
  Coefficient of correlation between the change from baseline in FEV1 with indacaterol after 1 month and the reversibility to salbutamol at screening

SECONDARY OUTCOMES:
Coefficient of correlation between VQ11 (an assessment of quality of life) and reversibility | 5 months
  Coefficient of correlation between the change from baseline in VQ11 with indacaterol after 5 months and the reversibility to salbutamol at screening

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (120):
- France (120):
  - Novartis Investigative Site, Ferolles-Attily, France
  - Novartis Investigative Site, Suresnes, France
  - Novartis Investigative Site, Vernon, France
  - Novartis Investigative Site, Abbeville
  - Novartis Investigative Site, Ajaccio
  - Novartis Investigative Site, Albi
  - Novartis Investigative Site, Amboise
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Angoulême
  - Novartis Investigative Site, Argenteuil
  - Novartis Investigative Site, Arles
  - Novartis Investigative Site, Armentières
  - Novartis Investigative Site, Aubergenville
  - Novartis Investigative Site, Bastia
  - Novartis Investigative Site, Beauvais
  - Novartis Investigative Site, Belfort
  - Novartis Investigative Site, Bergerac
  - Novartis Investigative Site, Bédarieux
  - Novartis Investigative Site, Béziers
  - Novartis Investigative Site, Blois
  - Novartis Investigative Site, Bois-Guillaume
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Boulogne-Billancourt
  - Novartis Investigative Site, Briançon
  - Novartis Investigative Site, Briey
  - Novartis Investigative Site, Cambrai
  - Novartis Investigative Site, Castelnau-le-Lez
  - Novartis Investigative Site, Ceret
  - Novartis Investigative Site, Chauny
  - Novartis Investigative Site, Châteaubriant
  - Novartis Investigative Site, Châteauroux
  - Novartis Investigative Site, Châtellerault
  - Novartis Investigative Site, Chelles
  - Novartis Investigative Site, Cherbourg Octeville
  - Novartis Investigative Site, Cholet
  - Novartis Investigative Site, Cognac
  - Novartis Investigative Site, Colmar
  - Novartis Investigative Site, Compiègne
  - Novartis Investigative Site, Dieulefit
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Dole
  - Novartis Investigative Site, Ermont
  - Novartis Investigative Site, Écully
  - Novartis Investigative Site, Forbach
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Grenoble Cédex 9
  - Novartis Investigative Site, Herblay-sur-Seine
  - Novartis Investigative Site, Hénin-Beaumont
  - Novartis Investigative Site, Ismer
  - Novartis Investigative Site, Jean de Verges
  - Novartis Investigative Site, L'Aigle
  - Novartis Investigative Site, La Chausse Saint Victor
  - Novartis Investigative Site, La Garde
  - Novartis Investigative Site, La Teste-de-Buch
  - Novartis Investigative Site, Le Cannet
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Le Perreux-sur-Marne
  - Novartis Investigative Site, Lens
  - Novartis Investigative Site, Libourne
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Lomme
  - Novartis Investigative Site, Lunel
  - Novartis Investigative Site, Lunéville
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Metz
  - Novartis Investigative Site, Molsheim
  - Novartis Investigative Site, Mont-de-Marsan
  - Novartis Investigative Site, Mont-Saint-Martin
  - Novartis Investigative Site, Montauban
  - Novartis Investigative Site, Montbéliard
  - Novartis Investigative Site, Montfermeil
  - Novartis Investigative Site, Montigny-lès-Metz
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Mulhouse
  - Novartis Investigative Site, Nancy
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Narbonne
  - Novartis Investigative Site, Nevers
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Obernai
  - Novartis Investigative Site, Ollioules
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Perpignan
  - Novartis Investigative Site, Péronne
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Quimper
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Roubaix
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Royan
  - Novartis Investigative Site, Saint-Gaudens
  - Novartis Investigative Site, Saint-Quentin
  - Novartis Investigative Site, Sainte-Feyre
  - Novartis Investigative Site, Saintes
  - Novartis Investigative Site, Salon-de-Provence
  - Novartis Investigative Site, Sceaux
  - Novartis Investigative Site, Sélestat
  - Novartis Investigative Site, Soissons
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Taden
  - Novartis Investigative Site, Thiais
  - Novartis Investigative Site, Thionville
  - Novartis Investigative Site, Thouars
  - Novartis Investigative Site, Toul
  - Novartis Investigative Site, Toulon
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Tulle
  - Novartis Investigative Site, Vandoeuvre Les Nancys
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
  - Novartis Investigative Site, Vesoul
  - Novartis Investigative Site, Vénissieux
  - Novartis Investigative Site, Vienne
  - Novartis Investigative Site, Villefranche-sur-Saône

REFERENCES:
- [Derived] Burgel PR, Le Gros V, Decuypere L, Bourdeix I, Perez T, Deslee G. Immediate salbutamol responsiveness does not predict long-term benefits of indacaterol in patients with chronic obstructive pulmonary disease. BMC Pulm Med. 2017 Jan 31;17(1):25. doi: 10.1186/s12890-017-0372-z. PMID 28143447